CLINICAL TRIAL: NCT06853743
Title: The NAD-HD Study: A Parallel-group, Phase 2, Double-blind Study to Investigate the Efficacy and Safety of Oral Nicotinamide Riboside Compared With Placebo in Participants Aged 18 to 80 Years With Huntington's Disease
Brief Title: The NAD-HD Study: A Study to Investigate Efficacy and Safety of Nicotinamide Riboside Compared With Placebo in Huntington's Disease
Acronym: NAD-HD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); South-Eastern Norway Regional Health Authority (Other); Klinbeforsk (Other); The Dam Foundation (Other); Elysium Health (Industry); NKS Olaviken Gerontopsychiatric Hospital (Other)
Responsible Party: Principal Investigator, Lasse Pihlstrøm, Senior Consultant and Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 803276; 2023209 (Other Grant/Funding Number: Clinical therapy research in the specialist health services (KLINBEFORSK), Norway)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Huntington Disease
Keywords: Huntington's disease; Nicotinamide riboside; Vitamin B3; NAD; Neuroprotection
MeSH Terms: conditions — Huntington Disease | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide riboside (Experimental): Nicotinamide riboside, 2 capsules of 500mg twice daily
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)
- Placebo (Placebo Comparator): Nicotinamide riboside, 2 capsules twice daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — Nicotinamide riboside, 2 capsules of 500mg taken twice daily for 2 years
  Arms: Nicotinamide riboside
Dietary Supplement: Placebo — Placebo, 2 capsules twice daily for 2 years
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if oral supplement of nicotinamide riboside (NR), a form of vitamin B3, slows disease progression in adults with Huntington's disease. It will also learn about the safety of nicotinamide riboside. The main questions it aims to answer are:

* Does NR slow progression of overall symptom burden in Huntington's disease?
* Does NR have an effect on any specific symptom domain in Huntington's disease?
* Does supplementation with NR cause side-effects or safety issues when used for 2 years in Huntington's disease?
* Does NR have an effect on selected blood, imaging, and oculomotor biomarkers in Huntington's disease?

Researchers will compare NR to a placebo (a look-alike substance that contains no active compound) to see if NR works to treat Huntington's disease.

Participants will:

* Take 2000mg NR or a placebo every day for 2 years
* Visit the clinic once every 6 months for clinical investigations and tests
* Undergo brain imaging at baseline and upon completion of the study period

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HD gene expansion carrier status with a diagnostic genetic test confirming ≥36 CAG-repeats in HTT.
* Clinically manifest HD with objective neurological signs corresponding to Diagnostic Confidence Level 4 based on the Total Motor Score of the UHDRS.
* Early or mid-stage disease corresponding to Shoulson-Fahn stage 1-340 and Total Functional Capacity (TFC) > 2.
* Ability to walk indoors unassisted or by the help of walking aids only as determined at screening and baseline visits.
* Ability to write and perform pen-and-paper tests (SDMT, SWRT, MoCA) and complete questionnaires (HADS-SIS, SF-12) included in the study protocol.
* Ability to follow up telephone appointments and reliably attend study visits independently or with the assistance of a reliable partner (family member, friend, or assistant).
* Ability to tolerate blood draws.
* Participants who are women of childbearing potential should use an approved method for highly effective birth control throughout the study intervention period
* Capable of giving signed informed consent

Exclusion Criteria:

* Presence of other co-morbid neurological or psychiatric disorders considered clinically significant by the investigator, including, but not limited to psychotic disorders, brain tumor or inflammatory neurological disease.
* Attempted suicide or active suicidal ideation within 12 months prior to screening.
* A history of alcohol or substance use within a 12 month period prior to the baseline visit, fulfilling criteria of dependence or abuse under the International Classification of Diseases (ICD-10) F10-F19 (not including tobacco dependence).
* Any malignancy within 5 years prior to screening (except basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated) or history of a previously treated malignant disorder > 5 years prior to screening with a remaining clinically significant recurrence risk.
* Established coronary artery disease or clinically significant cerebrovascular disease as deemed by the investigator.
* High age-specific cardiovascular risk as defined by the NORRISK2 algorithm based on smoking status, systolic blood pressure, serum total cholesterol and family history, modeled on the Norwegian population
* Any medical condition which, in the investigator's judgement, may preclude the subject's safe participation in the study, interfere with the ability to comply with study procedures or confound the interpretation of study results.
* Use of vitamin B3 supplements in any form or dose during the study or within 3 months prior to screening.
* Planned major surgery of any kind during the study period that is likely to affect clinical ratings, including, but not limited to, joint replacement and spinal surgery.
* Electroconvulsive therapy.
* Any medical therapy with known severe side effects that, in the investigator's judgement, may preclude the subject's safe participation in the study, interfere with the ability to comply with study procedures or confound the interpretation of study results.
* Any history of gene therapy exposure for the treatment of HD.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-18 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the composite Unified Huntington's Disease Rating Scale at 730 days | From baseline to the end of treatment at 730 days (2 years)
  The cUHDRS is a composite outcome measure comprised of motor, cognitive and global functional components. It is calculated as an equally weighted sum of Z-scores, with lower scores indicating greater clincial burden of HD symptoms.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | From baseline to the end of treatment at 730 days
  Adverse events will be defined and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) and reported for each study arm.
Change from Baseline in the Unified Huntington's Disease Total Motor Score at 730 days | From baseline to the end of treatment ao 730 days
  The Unified Huntington's Disease Total Motor Score is the sum of 30 items rated from 0 to 4 based on a clinical neurological assessment, where 0 is normal and 4 indicates the most severe motor deficit.
Change from Baseline in the Montreal Cognitive Assessment at 730 days | From baseline to the end of treatment at 730 days
  The Monteal Cognitive Assessment is a brief clinical test where results range from 0 to 30, and a higher score indicates better performance.
Change from baseline in the Hospital Anxiety and Depression Scale/Snaith Irritability Scale (HADS-SIS) at 730 days | From baseline to the end of treatment at 730 days
  The Hospital Anxiety and Depression Scale/Snaith Irritability Scale (HADS-SIS) is a questionnaire completed by the participant with 22 questions,. Replies to each question are scored from 0 to 4, where 0 is normal and 4 is the most severe symptom

OTHER OUTCOMES:
Progression of Caudate Atrophy | From baseline to the end of treatment at 730 days
  Change in the volume of the caudate nucleus as measured by volumetric MRI
Change in Brain Metabolic Patterns | From baseline to the end of treatment at 730 days
  Change in glucose metabolic pattern as measured by fluorodeoxyglucose positron emission tomography (FDG-PET)
Change in Biomarker of Neuronal Damage | From baseline to the end of study treatment at 730 days
  Change in serum levels of neurofilament light chain (NfL)
Change in Markers of Inflammation | From baseline to the end of study treatment at 730 days
  Change in serum levels of selected inflammatory cytokines
Progression of Eye Movement Abnormalities | From baseline to the end of study treatment at 730 days
  Change in selected measures of saccades and fixation recorded by digital eye-tracking
Change in Health-Related Quality of Life | From baseline to the end of study treatment at 730 days
  Change in in health-related quality of life as measured by the 12-item Short Form Survey v2 (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Pihlstrøm, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway